CLINICAL TRIAL: NCT00578266
Title: Allogeneic Stem Cell Transplantation for Patients With Severe Aplastic Anemia, Using Matched Unrelated Donors and Mismatched Related Donors
Brief Title: Allogeneic Stem Cell Transplantation for Patients With Severe Aplastic Anemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Shakila Khan, MD, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-006216
Record Dates: First submitted 2007-12-17; First posted 2007-12-21 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Anemia, Aplastic
Keywords: Severe Aplastic Anemia (SAA); Transplant for Severe Aplastic Anemia (SAA)
MeSH Terms: conditions — Anemia, Aplastic | interventions — Cyclophosphamide; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- No Arms (Other)
  Interventions: Drug: Cyclophosphamide,Campath IH and TBI

INTERVENTIONS:
Drug: Cyclophosphamide,Campath IH and TBI — DAY 5 TREATMENT
  * 6 5 CYTOXAN 50 mg/kg WITH MESNA
  * 5 CYTOXAN 50 mg/kg WITH MESNA;
  * 4 CYTOXAN 50 mg/kgWITH MESNA; CAMPATH 3-10 mg
  * 3 CYTOXAN 50 mg/kg WITH MESNA; CAMPATH;
  * 2 TBI; CAMPATH; TACROLIMUS
  * 1 TBI (second fraction); CAMPATH (am) 0 STEM CELL INFUSION (pm)

SUMMARY:
For patients with severe aplastic anemia (SAA) who have failed to respond to immunosuppressive therapy and lack an HLA identical family member, our objectives are to make an initial assessment of the safety and efficacy of allogenic stem cell transplantation from either a matched unrelated donor or a mismatched reacted donor using the conditioning regimen of Cytoxan, reduced total body irradiation (TBI) and Campath IH. The principle measures of safety and efficacy will be :

1. Patient survival probability at 100 days, 1 year and 2 years.
2. Incidence of graft versus host disease (GVHD), as well as incidence of acute GVHD and chronic GVHD within 6 months and 2 years.
3. Engraftment at 6 months, 1 year and 2 years

DETAILED DESCRIPTION:
The objective of this trial is to make an initial assessment for this new treatment regimen and to show it is equal or superior to the current standard practice. With this initial assessment be hope to gain information suggesting further study of this regimen or discontinuation of this regimen before exposing large numbers of patients to this new treatment option. We also will gain experience with this new regimen giving insights as to possible modifications in dosing and monitoring and selection of patients for future treatment in case of positive results. For this initial study we plan to enroll up to 24 patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of SAA based on bone marrow aspirate and biopsy results. Failure to respond to immunosuppressive therapy and/or lack of an HLA identical family member.
* A 10/10 or 9/10 HLA matched unrelated donor or a 9/10 matched related donor available after high resolution typing.

Exclusion Criteria:

* Patients with Aplastic anemia and active infection must be treated to maximally resolve this problem before beginning the conditioning regimen.
* HIV seropositive patients
* Patients who have clonal cytogenetic abnormalities or a myelodysplastic syndrome.
* Patient greater than 60 years of age.
* Women who are pregnant or nursing.
* Patients with active hepatitis
* Patients with severe cardiac dysfunction defined as shortening fraction <25%.
* Patients with severe renal dysfunction defined as creatinine clearance <40ml/mim/1.73m2.
* Patient with severe pulmonary dysfunction with FEV1, FVC and DLCO 40% of predicted or 3 SD below normal.

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2007-02; Primary Completion 2016-08-16 (Actual); Study Completion 2016-08-16 (Actual)

PRIMARY OUTCOMES:
1. Engraftment at 6 months, 1 year and 2 years 2.Incidence of graft versus host disease (GVHD), as well as incidence of acute GVHD and chronic GVHD within 6 months and 2 years | 2 years

SECONDARY OUTCOMES:
Patient survival probability at 100 days, 1 year and 2 years. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Shakila P. Khan, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States